CLINICAL TRIAL: NCT05872607
Title: The Quantitative Study of the Habenula Based on Multi-channel Cascaded Neural Network and the Establishment of the Prediction Model of the Curative Effect in Patients With Depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: zlei19810830
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-02

CONDITIONS: Depression
Keywords: Depression; Habenula; Convolution neural network; Segmentation; Curative effect prediction
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Depression is the second leading cause of disease burden in our country. It has serious effects on the physical and mental health of human beings, and about 30% of patients with depression are unresponsive or respond poorly to antidepressant treatment. Clinical practice is in a tough position of wanting objective measures of assessing depression. The applicant and her team have devoted many years to the basic and clinical research on habenular nucleus (Hb) accumulating a significant amount of experience from animal experiments and patients' magnetic resonance (MR) studies. These studies have demonstrated that the habenular nucleus is the key target area that is responsible for the pathophysiological changes in depression as well as its treatment. Small volumes and unsatisfactory contrast have been knotty problems in the MR imaging of Hb. In addition, time-consuming manual segmentation and lack of quantitative standards in conventional studies has impeded the advancement of Hb research. Fortunately, the development of high-resolution multi-parametric quantitative MR imaging and the extensive use of artificial intelligence (AI) technology in medical imaging can just provide powerful support for the imaging, segmentation and quantification of Hb. This project proposes to use high resolution MR anatomy of Hb combined with multimodal fusion to 1) construct a model for automatic 3D segmentation of Hb MR images based on the densely connected multichannel dilated convolutional neural networks; 2) sift out the quantitative imaging signatures related to the antidepressants' efficacy using the radiomics methodology, and in combination with clinical information, construct an individualized prediction model for treatment efficacy.

Overall, this study focuses on the translation of basic research to clinical application in the hope of providing quantifiable objective imaging markers in clinical practice, facilitating clinical decision-making and bringing about individualized precise diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Premiere depressed patients

Exclusion Criteria:

* Drug therapy modality change、Incomplete MR image data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Premiere depressed patients
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Multimodal MR data of habenula | Baseline (Before medication)
  To extract high-dimensional features of multimodal image data including MP2RAGE, T1MAP, T2 SPACE, DIR, QSM, T2 *

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China